CLINICAL TRIAL: NCT02359825
Title: Nerve Repair Using Hydrophilic Polymers to Promote Immediate Fusion of Severed Axons and Swift Return of Function
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Wesley Thayer, MD, PHD, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 191655
Record Dates: First submitted 2015-02-04; First posted 2015-02-10 (Estimated); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Peripheral Nerve Injury
MeSH Terms: conditions — Peripheral Nerve Injuries | interventions — Polyethylene Glycols

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- standard epineural repair <24 hours (No Intervention): epineural repair following treatment with standard epineural repair alone in sensory nerve injuries in the upper extremity in short-term acute injuries (repaired <24 hours after injury); no medication used
- standard epineural repair >24 - 72 hours (No Intervention): epineural repair following irrigation with standard epineural repair alone in sensory nerve injuries in the upper extremity in short-term chronic injuries (>24-<72 hours after injury); no medication used
- epineural repair with autografting within 48 hours (No Intervention): epineural repair with auto grafting within 48 hours; no medication used
- epineural repair <24 hours using PEG (Experimental): epineural repair following treatment with standard epineural repair using PEG in sensory nerve injuries in the upper extremity in short-term acute injuries (repaired <24 hours after injury); PEG is used during the surgical procedure
  Interventions: Drug: Polyethylene glycol (PEG)
- epineural repair >24 but <72 hours using PEG (Experimental): epineural repair following treatment with standard epineural repair using PEG in sensory nerve injuries in the upper extremity in short-term acute injuries (repaired >24 hours but < 72 hours after injury); PEG is used during the surgical procedure
  Interventions: Drug: Polyethylene glycol (PEG)
- epineural repair with autografting within 48 hours, using PEG (Experimental): epineural repair with auto grafting within 48 hours
  Interventions: Drug: Polyethylene glycol (PEG)

INTERVENTIONS:
Drug: Polyethylene glycol (PEG) — For the control groups, epineural repair or interposition grafting will be undertaken in the standard end-to-end fashion using interrupted nylon suture after irrigation of the wound with normal saline as deemed necessary by the operating surgeon. For the experimental group, the nerve(s) will be repaired using standard suture neurorrhaphy techniques and a 149.25 mM (50%) solution of PEG 3.35 kD in sterile water will then be irrigated onto the neurorrhaphy site for one minute. Following this, the approximated nerve ends will be irrigated with sterile water gently for 2 minutes. All wounds will be closed in the fashion deemed appropriate by the operating surgeon.
  Other Names: PEG
  Arms: epineural repair <24 hours using PEG; epineural repair >24 but <72 hours using PEG; epineural repair with autografting within 48 hours, using PEG

SUMMARY:
Current strategies for peripheral nerve repair are severely limited. Even with current techniques, it can take months for regenerating axons to reach denervated target tissues when injuries are proximally located. This inability to rapidly restore the loss of function after axonal injury continues to produce poor clinical outcomes. The investigators propose testing the efficacy and safety of a combination therapy: polyethylene glycol (PEG) assisted axonal fusion technique to repair peripheral nerve injuries in humans.

DETAILED DESCRIPTION:
Our own preclinical animal studies have been designed to take advantage of PEG. We have used the fusogenic properties of PEG and this has allowed us to demonstrate a rapid and decisive electrophysiological recovery of either crushed or completely severed sciatic nerves in a commonly accepted mammalian model for peripheral nerve injury (Bittner et al JSR 2012).

Recently, we modified previously published mammalian techniques. Our goal was to eliminate laboratory solutions that have not been approved for use in humans and replace them with readily available reagents commonly used in clinical applications. PEG is commercially available in many molecular formulations and our earlier experiments with PEG having a molecular weight of 2 kD. Unfortunately, this molecular weight is not approved by the Food and Drug Administration (FDA) for human usage. In our more recent preclinical studies, we have demonstrated that PEG 3.35 kD, the main ingredient in the commonly used cathartic known as MiraLAX© (MERCK; Whitehouse Station, NJ), actually generates superior fusion over PEG 2KD in a cut nerve model. Thus the clinical trial that forms the basis of this proposal was developed with the FDA approved 3.35 kD PEG and these other two FDA approved solutions.

Additional studies in our complex nerve injury model have also demonstrated that the repair does not have to be performed immediately after nerve injury. Epineural repair with PEG 3.35 kD treatment can be performed up to 24hrs after injury and postoperative CAPs are obtained in all PEG 3.35 kD treated animals (n=3, data not shown). The remarkable finding is that in the 24-hour injury model, PEG significantly improves behavioral outcome measured at 72 hours postoperatively.

Based on the published reports and our own in vivo studies, we demonstrate that PEG based repair can restore CAPs immediately and improve functional recovery significantly post injury. These preclinical findings suggest that we can offer a novel therapy to test in humans who have experienced complete transection of a peripheral nerve. Patient risk is minimized as we have optimized the PEG facilitated fusion technique to utilize commonly used FDA approved drugs, solutions and electrolytes to augment standard neurorrhaphy techniques. The experimental protocol entails 100% transection injury to a peripheral nerve followed by a standard neurorrhaphy. The repair is then irrigated gently with PEG for two minutes and sterile water in standard fashion is used to wash away the PEG.

The most likely scenarios, that explain rapid compound action potential (CAP) restoration, are the rapid restoration of cytoplasmic flow within the nerves, the rapid ability of membranes to depolarize and possibly the prevention of Wallerian degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a Sunderland Class 5 traumatic neuropathy (transection injury) of a digital nerve in the upper extremity
* candidates for immediate operative repair (Arm 1);
* injury proceeding repair no longer than 72 hours; and
* repair within 48 hours of injury that require nerve grafting;
* N0 significant medical comorbidities precluding immediate repair;
* willing to comply with all aspects of the treatment and evaluation schedule over a 12 months period.

We plan to include subjects who have peripheral nerve injuries that are complicated by significant vascular or orthopedic damage.

Exclusion Criteria:

* Patients will be excluded from enrollment if their injuries exhibit gross contamination, in circumstances where soft tissue coverage is inadequate, or when staged repair is planned.
* We will also exclude patients that are diabetic, have been diagnosed with a neuromuscular disease, or are undergoing chemotherapy, radiation therapy, or other treatments known to affect the growth of the neural and vascular system.
* We will exclude all patients currently enrolled in another investigational study or those who are unlikely to complete the normal regime of occupational therapy. Individuals will be excluded from participation if their time of injury falls outside study parameters.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-09-19 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
return of nerve function as measured by (Medical Research Council Classificatoin (MRCC) | 12 months
  Medical Research Council Classificatoin (MRCC)

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Thayer, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No